CLINICAL TRIAL: NCT02534467
Title: Montelukast as Adjunct Treatment in Children With Atopic Dermatitis
Brief Title: Does Treatment With Montelukast Improve Symptoms of Atopic Dermatitis in Children?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 35095A
Record Dates: First submitted 2015-08-13; First posted 2015-08-27 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — montelukast

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montelukast-Standard (Experimental): 8 weeks of montelukast and standard therapy crossing over to 8 weeks of only standard therapy
  Interventions: Drug: Montelukast
- Standard-Montelukast (Active Comparator): 8 weeks of standard therapy only crossing over to 8 weeks of montelukast and standard therapy
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — daily dose according to age for 8 weeks out of 16 weeks of assessment
  Other Names: Apo-Montelukast, Singulair

SUMMARY:
An open-label (outcome assessor blinded) prospective crossover cohort study of children 6-16 years assessing effects of Montelukast on moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
An open-label, prospective cohort study with two arms over 16 weeks comprising 8 weeks of treatment with montelukast and 8 weeks without treatment of montelukast. All patients will be followed from recruitment to the study end date.

Study Population 62 patients aged 6-16 years old with moderate to severe atopic dermatitis recruited from the Royal Children's Hospital and Box Hill Hospital dermatology clinics having already previously received eczema education (SCORAD >25) Study Product Oral tablet montelukast Dose Regimen For patients 6-8 years old - 4mg montelukast once daily For patients 9-13 years old - 5mg montelukast once daily For patients 14-16 years old - 10mg montelukast once daily Evaluation Criteria Primary objective measurement: mean change in SCORAD index at 8 weeks Patients will be randomized into 2 arms: Arm 1 treated with montelukast therapy over 8 weeks followed by no montelukast therapy for 8 weeks. Arm 2 followed for 8 weeks without montelukast therapy followed by 8 weeks with montelukast therapy.

Assessment Schedule Clinical assessment will be conducted at baseline (week 0), and reviewed every 4 weeks over 16 weeks with a safety follow-up visit 2 weeks after the treatment ends (week 18). At the first clinic visit, demographic data, medical history and baseline SCORAD and cDLQI will be recorded. cDLQI will be completed by the participants. Participants with SCORAD <25 are considered to have mild disease and will not be included in the study. Suitable participants will be prescribed oral montelukast as an adjunct to their standard topical therapy (corticosteroids, emollients) or immunosuppressive therapy. Adverse effects, SCORAD (assessed by a blinded assessor) and cDLQI will be assessed at each review.

Data will be analyzed based on intention-to-treat. Paired data on SCORAD and cDLQI will be analyzed. A p value <0.05 will be considered statistically significant. A 30% improvement in SCORAD and cDLQI scores will be considered clinically significant.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 6-16 years old with moderate to severe atopic dermatitis (SCORAD >25) despite topical therapy (corticosteroids and emollients) for at least 2 months Patients aged 6-16 years old with moderate to severe atopic dermatitis (SCORAD >25) despite immunosuppressive therapy (azathioprine, cyclosporine, methotrexate) for at least 2 months

Exclusion Criteria:

- Patients with mild atopic dermatitis (SCORAD <25) Patients who have received phototherapy in the past 8 weeks Patients with history of sensitivity to leukotriene receptor antagonists

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Change in SCORAD Scoring Atopic Dermatitis index (Units on a scale) | at 8 weeks
  assessed by blinded assessor

SECONDARY OUTCOMES:
Change in SCORAD Scoring Atopic Dermatitis index (Units on a scale) | at 4 weeks
  assessed by a blinded assessor
Change in children's Dermatology Life Quality Index cDLQI (Units on a scale) | at 8 weeks
Change in children's Dermatology Life Quality Index cDLQI (Units on a scale) | at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John C Su, FRACP, FACD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- The Royal Children's Hospital, Parkville, Victoria, Australia